CLINICAL TRIAL: NCT05934383
Title: Safety and Efficacy of Ultrasound Renal Denervation in Kidney Transplantation Patients With Uncontrolled Hypertension: the RESTART Study
Brief Title: Safety and Efficacy of Ultrasound Renal Denervation in Kidney Transplantation Patients With Uncontrolled Hypertension
Acronym: RESTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ReCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Joost Daemen, Interventional cardiologist, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTART - renal denervation
Record Dates: First submitted 2023-06-25; First posted 2023-07-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Kidney Transplantation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renal sympathetic denervation (Experimental)
  Interventions: Device: Paradise® ultrasound renal denervation system.

INTERVENTIONS:
Device: Paradise® ultrasound renal denervation system. — Bilateral renal sympathetic denervation of the native kidneys using the Paradise® ultrasound renal denervation system.

SUMMARY:
This prospective, single-arm, interventional study is designed to assess the short-term and long-term safety and efficacy of bilateral ultrasound renal sympathetic denervation (RDN) of the native kidneys in renal transplant patients with uncontrolled hypertension.

Objectives:

* To assess the short-term and long-term changes in ambulatory and office blood pressure (BP) following native kidney RDN in renal transplant patients
* To assess the long-term safety of native kidney RDN in renal transplant patients
* To assess the short-term and long-term change in antihypertensive drug prescriptions following native kidney RDN in renal transplant patients
* To assess the short-term and long-term change in adherence to antihypertensive drugs following native kidney RDN in renal transplant patients

DETAILED DESCRIPTION:
The RESTART study is an investigator-initiated, prospective, single-center, single-arm interventional study investigating the safety and efficacy of bilateral native kidney RDN in 40 renal transplant patients with uncontrolled hypertension despite antihypertensive medication (or with a documented intolerance to antihypertensive drugs).

Previously, RDN demonstrated to safely reduce BP as compared to sham-control in multiple randomized clinical trials, both in patients with and without concomitant antihypertensive medication. Up until now, patients with a history of renal failure or kidney transplantation have been excluded from these studies. As the pathophysiology of hypertension is considered different in hypertensive renal transplant patients as compared to the previously studied populations (without kidney transplantation), the effect of native kidney RDN in hypertensive patients with a history of kidney transplantation remains unknown. The current study aims to provide novel insights on the safety and efficacy of RDN in this particular population. Adjustment for routine therapy adherence will also be performed as this proved to be an important confounding factor in previous research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Kidney transplantation ≥ 12 months ago with stable immunosuppressive drug treatment
* Estimated Glomerular Filtration Rate (eGFR) ≥ 40 ml/min/1.73m2
* Office systolic BP ≥ 140 mmHg and a mean 24-hour ambulatory systolic BP ≥ 130 mmHg at screening
* Antihypertensive medication regimen:

  * Stable regimen of at least two antihypertensive drugs of different classes, including a diuretic (defined a thiazide diuretic, loop diuretic or mineralocorticoid receptor antagonist), for at least three months, or
  * Documented intolerance to three classes of antihypertensive drugs, and
  * A change in antihypertensive drug regimen is not anticipated within the oncoming three months.
* Patient is willing and able to provide written informed consent

Exclusion Criteria:

* Native renal artery anatomy not eligible for RDN, defined as at least one of the following conditions:

  * History of renal artery stenting or angioplasty
  * History of renal denervation
  * History of kidney tumors
  * Renal artery diameter < 3 mm or > 8 mm
  * Renal artery length < 20 mm
  * Fibromuscular disease (FMD) of the native renal arteries
  * Renal artery aneurysm
  * Renal artery stenosis > 30%
* Presence of a remnant transplant kidney after re-transplantation or absence of native kidneys
* Solitary native kidney
* History of intravenous contrast dye allergy or nephropathy
* Iliac/femoral artery stenosis precluding insertion of the Paradise catheter
* Uncorrected, treatable secondary cause of hypertension
* Pregnancy
* Life expectancy < one year at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy: change in mean 24-hour ambulatory systolic blood pressure | Baseline vs. 3-month follow-up
Safety: occurrence of the composite endpoint | Baseline vs. 3-month follow-up
  Consisting of (whichever occurs first):
  * All-cause mortality
  * New onset (acute) end-stage renal disease (eGFR< 15 mL/min/m2 or need for renal replacement therapy)
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation requiring an invasive intervention
  * Renal artery dissection requiring an invasive intervention
  * Major vascular complications
  * Hospitalization for hypertensive or hypotensive crisis

SECONDARY OUTCOMES:
Efficacy: change in mean 24-hour ambulatory diastolic blood pressure | Baseline vs. 3-month follow-up
Efficacy: change in daytime ambulatory systolic and diastolic blood pressure | Baseline vs. 3-month follow-up
Efficacy: change in nighttime ambulatory systolic and diastolic blood pressure | Baseline vs. 3-month follow-up
Efficacy: change in office systolic and diastolic blood pressure | Baseline vs. 3-month follow-up
Efficacy: changes in ambulatory (mean 24-hour, daytime, nighttime) systolic and diastolic blood pressure | Baseline vs. 3-month follow-up
  In a subpopulation of patients with an equal level of therapy adherence at both timepoints
Efficacy: changes in office systolic and diastolic blood pressure | Baseline vs. 3-month follow-up
  In a subpopulation of patients with an equal level of therapy adherence at both timepoints
Efficacy: changes in the number of prescribed defined daily dosages and number of classes of antihypertensive drugs | Baseline vs. 3-month follow-up
Efficacy: change in the percentage therapy adherence | Baseline vs. 3-month follow-up
  The percentage adherence will be calculated as the proportion of drugs that could be detected using dried blood spot testing out of all drugs prescribed to the patient at the time of the testing.
Efficacy: annual changes in ambulatory (mean 24-hour, daytime, nighttime) systolic and diastolic blood pressure | Baseline up until and including 5-year follow-up
Efficacy: annual changes in office systolic and diastolic blood pressure | Baseline up until and including 5-year follow-up
Efficacy: annual changes in in the number of prescribed defined daily dosages and number of classes of antihypertensive drugs | Baseline up until and including 5-year follow-up
Efficacy: annual change in the percentage therapy adherence | Baseline up until and including 5-year follow-up
  The percentage adherence will be calculated as the proportion of drugs that could be detected using dried blood spot testing out of all drugs prescribed to the patient at the time of the testing.
Safety: the number of patients in whom no successful bilateral renal denervation procedure can be performed | Periprocedural
  E.g. due to anatomical difficulties
Safety: change in renal function (estimated Glomerular Filtration Rate) | Baseline vs. 3-month follow-up
Safety: change in renal function (urine protein/creatinine ratio) | Baseline vs. 3-month follow-up
Safety: occurrence of the individual components of the primary safety outcome | Baseline up until and including 5-year follow-up
  * All-cause mortality
  * New onset (acute) end-stage renal disease (eGFR< 15 mL/min/m2 or need for renal replacement therapy)
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation requiring an invasive intervention
  * Renal artery dissection requiring an invasive intervention
  * Major vascular complications
  * Hospitalization for hypertensive or hypotensive crisis
Safety: occurrence of any major adverse cardiovascular and cerebrovascular event (MACCE) | Baseline up until and including 5-year follow-up
  Including myocardial infarction, coronary revascularization, stroke and cardiovascular mortality
Safety: occurrence of the individual components of major adverse cardiovascular and cerebrovascular event (MACCE) | Baseline up until and including 5-year follow-up
  Including myocardial infarction, coronary revascularization, stroke and cardiovascular mortality
Safety: annual change in renal function (estimated Glomerular Filtration Rate) | Baseline up until and including 5-year follow-up
Safety: annual change in renal function (urine protein/creatinine ratio) | Baseline up until and including 5-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands